CLINICAL TRIAL: NCT01832350
Title: Clinical Protocol of a Prospective, Open-label Study to Assess the Safety and Efficacy of Nuedexta (Dextromethorphan/Quinidine) in the Treatment of Pseudobulbar Affect (PBA) in Patients With Alzheimer's Disease
Brief Title: Nuedexta in the Treatment of Pseudobulbar Affect in Patients With Alzheimer's Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor decided to stop study early
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Collaborators: Avanir Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AVP923
Record Dates: First submitted 2013-04-09; First posted 2013-04-16 (Estimated); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Alzheimer's Disease; Pseudobulbar Affect (PBA)
MeSH Terms: conditions — Alzheimer Disease | interventions — dextromethorphan - quinidine combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nuedexta (20/10) (Experimental): Drug: Nuedexta (20/10) administered orally, two times a day (every 12 hours), during a 26-week period.
  Interventions: Drug: Nuedexta (20/10)

INTERVENTIONS:
Drug: Nuedexta (20/10) — Drug: Nuedexta (20/10) administered orally, two times a day, every 12 hours, during a 26-week period.
  Other Names: Dextromethorphan/Quinidine

SUMMARY:
The primary objective of this study is to test the hypothesis that Nuedexta (20/10) administered orally will reduce Pseudobulbar Affect (PBA) frequency and severity (CNS-Lability Scale and PLACS), with satisfactory safety and high tolerability in patients with Alzheimer's Disease (AD). The primary objective will be evaluated using a study endpoint at 1, 13, 26 weeks after initiation of treatment. The secondary objective of this study is to evaluate the benefit of treatment with Nuedexta (20/10) on cognition and functionality as demonstrated in the Rey Auditory Verbal Learning Test (RAVLT), Trail making A and B, Wechsler Memory Scale (WMS) logical memory and delayed recall, Controlled Oral Word Association (COWA), Clinical Dementia Rating (CDR), Neuropsychiatric Inventory (NPI), Alzheimer's Disease Cooperative Study Activities of Daily Living Inventory (ADCSADL) and the 11-item Alzheimer's Disease Assessment Scale-Cognitive subscore (ADAS-Cog11).

ELIGIBILITY:
Inclusion Criteria:

* Male/female 55 to 90 years, inclusive.
* Meets National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association criteria for probable AD.
* Modified Hachinski Ischemia Scale score of ≤4.
* Folstein Mini Mental State Exam score 16-26 at Visit 1.
* Geriatric Depression Scale score ≤6. For patient with history of depression, he/she have been on steady dose of anti-depressant for at least 3 months.
* Clinical history and relevant symptoms of Pseudobulbar Affect.
* Center for Neurologic Study-Lability Scale score at baseline ≥13.
* Stable hematologic, hepatic, and renal function, with no clinically significant symptoms, and with clinical laboratory results (CBC, clinical chemistry, and urinalysis) up to 1-fold higher than upper limit of normal range.
* Resting respiratory rate 12-20/minute.
* MRI or CT scan within past 12 months; no findings inconsistent with diagnosis of AD.
* ECG (within 4 weeks prior to entry)with no evidence of clinically significant abnormalities.
* Concurrent treatment with an acetylcholinesterase inhibitor or memantine allowed; must be on stable dose at least 2 months before screening. Dosing must remain stable throughout the study.
* Use of SSRI's allowed. Must have used for 3 months prior to study entry; dose must remain unchanged during course of study.
* No current symptoms of depressive disorder.
* Score of 19 or lower in the Beck Depression Inventory.
* Agrees to use no prohibited medications during study.

Exclusion Criteria:

* Has current serious or unstable illnesses that, in investigator's opinion, could interfere with analysis of safety and efficacy data; has life expectancy <2 years.
* No reliable caregiver in frequent contact with patient (at least 10 hours/week.
* Current or prior history of major psychiatric disturbance.
* Have been in other clinical study within 30 days of entry.
* Score of 20 or higher in Beck Depression Inventory.
* Multiple episodes of head trauma, history within last year of serious infectious disease affecting the brain, head trauma resulting in protracted loss of consciousness, or myasthenia gravis.
* Within the last 5 years, history of a primary or recurrent malignant disease.
* Known sensitivity to quinidine or dextromethorphan.
* History of human immunodeficiency virus, multiple or severe drug allergies, or severe post-treatment hypersensitivity reactions.
* History of chronic alcohol or drug abuse/dependence within the past 5 years.
* Judged by investigator to be at serious risk for suicide.
* Has a recent or current lab result indicating clinically significant lab abnormality.
* At Visit 1 has ALT/SGPT values ≥2 times upper limit of normal (ULN); AST/SGOT values ≥3 times the ULN; total bilirubin values ≥2 times the ULN.
* Resting diurnal oxygen saturation <95%.
* Received dextromethorphan and quinidine within previous 6 months.
* Hypotension (systolic BP <100 mm Hg); postural syncope; unexplained syncope.
* Used medications that affect the CNS (except for AD) for less than 4 weeks.
* On disallowed concomitant medications.
* Experiencing acute exacerbation of underlying neurological disorder within previous 2 months.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-08-28 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
reduction of PBA frequency | 1, 13, and 26 weeks after initiation of treatment

SECONDARY OUTCOMES:
reduction of PBA severity | 1, 13, and 26 weeks after initiation of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jiong Shi, MD, PhD, Principal Investigator — Barrow Neurological Institute, St. Joseph's Hospital and Medical Center, Phoenix AZ
Locations (1):
- Barrow Neurological Institute, Phoenix, Arizona, United States

REFERENCES:
- [Background] Schiffer R, Pope LE. Review of pseudobulbar affect including a novel and potential therapy. J Neuropsychiatry Clin Neurosci. 2005 Fall;17(4):447-54. doi: 10.1176/jnp.17.4.447. PMID 16387982
- [Background] Green RL. Regulation of Affect. Semin Clin Neuropsychiatry. 1998 Jul;3(3):195-200. PMID 10085207
- [Background] Lieberman A, Benson DF. Control of emotional expression in pseudobulbar palsy. A personal experience. Arch Neurol. 1977 Nov;34(11):717-9. doi: 10.1001/archneur.1977.00500230087017. PMID 911237
- [Background] Starkstein SE, Migliorelli R, Teson A, Petracca G, Chemerinsky E, Manes F, Leiguarda R. Prevalence and clinical correlates of pathological affective display in Alzheimer's disease. J Neurol Neurosurg Psychiatry. 1995 Jul;59(1):55-60. doi: 10.1136/jnnp.59.1.55. PMID 7608711
- [Background] Tanaka M, Sumitsuji N. Electromyographic study of facial expressions during pathological laughing and crying. Electromyogr Clin Neurophysiol. 1991 Oct-Nov;31(7):399-406. PMID 1748077
- [Background] Pioro EP, Brooks BR, Cummings J, Schiffer R, Thisted RA, Wynn D, Hepner A, Kaye R; Safety, Tolerability, and Efficacy Results Trial of AVP-923 in PBA Investigators. Dextromethorphan plus ultra low-dose quinidine reduces pseudobulbar affect. Ann Neurol. 2010 Nov;68(5):693-702. doi: 10.1002/ana.22093. PMID 20839238
- [Background] Strowd RE, Cartwright MS, Okun MS, Haq I, Siddiqui MS. Pseudobulbar affect: prevalence and quality of life impact in movement disorders. J Neurol. 2010 Aug;257(8):1382-7. doi: 10.1007/s00415-010-5550-3. Epub 2010 Apr 8. PMID 20376475
- [Background] Wolf JK, Santana HB, Thorpy M. Treatment of "emotional incontinence" with levodopa. Neurology. 1979 Oct;29(10):1435-6. doi: 10.1212/wnl.29.10.1435-b. No abstract available. PMID 573397